CLINICAL TRIAL: NCT05776758
Title: Neoadjuvant Chemotherapy Plus Cystectomy vs Cystectomy Alone for cT0 Muscle-invasive Bladder Cancer After Maximal TURBt: Multicentre Prospective Randomized Controlled Trial
Brief Title: Role of NAC in cT0 Muscle-invasive Bladder Cancer After Maximal TURBt
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Giuseppe SImone, MD, PhD, Chief of Urology, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RS1779/22(2738)
Record Dates: First submitted 2023-01-31; First posted 2023-03-20 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Muscle-Invasive Bladder Carcinoma; Chemotherapy Effect; Surgery
Keywords: Bladder cancer; Muscle-invasive bladder cancer; Radical cystectomy; Survival outcomes
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAC+RC (Experimental): cisplatin-based neoadjuvant chemotherapy plus radical cystectomy
  Interventions: Drug: cisplatin based neoadjuvant chemotherapy; Procedure: Radical cystectomy alone
- RC alone (Active Comparator): radical cystectomy alone
  Interventions: Procedure: Radical cystectomy alone

INTERVENTIONS:
Drug: cisplatin based neoadjuvant chemotherapy — cisplatin based neoadjuvant chemotherapy
  Arms: NAC+RC
Procedure: Radical cystectomy alone — RC alone

SUMMARY:
This prospective randomized controlled trial (RCT) is designed to provide high level evidence describing the non-inferiority of radical cystectomy (RC) alone versus neoadjuvant chemotherapy (NAC) plus RC on survival outcomes of patients with a diagnostic transurethral resection of bladder tumor (TURBt) of non-metastatic muscle invasive bladder cancer (MIBC) (T2-T4 N0 M0) and non-radiologic or endoscopic residual tumor after a maximal TURBt (cT0). Our hypothesis is that performing NAC in the absence of residual disease, after a maximal TURBt, has no survival benefit over performing an early cystectomy. Since no downstaging could be achieved in patients with no residual tumor into the bladder, the benefits of neoadjuvant chemotherapy in this setting could be not significant and it might turn into unnecessary toxicity and a substantial delay to surgical treatment.

DETAILED DESCRIPTION:
Radical Cystectomy (RC) is considered the reference option for treatment of urothelial muscle invasive bladder cancer (MIBC). However, RC alone has been reported 5-year survival in about 50% of patients. Therefore, to improve survival outcomes in patients with non-metastatic MIBC, cisplatin-based neoadjuvant chemotherapy (NAC) has been introduced. On the one hand, major tolerability, higher patient compliance and lower burden of micrometastatic disease are listed as potential advantages of administering NAC before planned definitive surgery. Several phase III randomized controlled trials (RCTs) reported the potential survival benefit of NAC administration.

Moreover, the updated analysis of a large phase III RCT, globally including all patients with muscle invasive bladder cancer from T2 to T4, regardless of post transurethral resection of bladder tumor (TURBt) tumor volume, with a median follow-up of 8-yrs confirmed previous results providing additional findings:

* 16% reduction in mortality risk;
* improvement in 10-yr survival from 30% to 36% with NAC;
* Benefit with regard to distant metastases;
* the addition of NAC provided no benefit for locoregional control and locoregional disease free survival (DFS).

On the other hand, the possibility to predict patients' sensitivity to chemotherapy is still limited. Therefore, the delay in performing RC and the theoretical impact of NAC on surgical morbidity are considered significant limitations to a routine administration of neoadjuvant treatments. As a result, it is growing the interest at improving selection clinical criteria to identify the ideal candidates to NAC, in order to obtain the maximal survival benefit of NAC, minimizing its possible disadvantages. Reliable predictive markers and molecular tumour profiling might guide the use of NAC in the future, but nowadays they are not currently used in clinical practice.

Despite the evidence supporting the use of NAC, its routine administration is still limited. The risk of unresponse after NAC, with the consequent delay in surgical treatment, and the possible impact on surgical morbidity after RC, are the major limitations to the wide administration of NAC. Previous evidences supported the use of NAC in patients with T2 to T4a BCa, regardless of tumor volume at the time of NAC. It is growing the interest on a tailored approach to treat genitourinary cancer, therefore it is needed much more efforts to select which patient will benefit most from NAC rather than an early RC. To answer this question, it is needed to selectively perform RCTs aiming to test specific treatments in equally specific patients. The primary objective of the trial is to demonstrate the non-inferiority of RC alone versus NAC plus RC on survival outcomes of patients with a diagnostic TURBt of non-metastatic muscle invasive bladder cancer (MIBC) (T2-T4 N0 M0) and non-radiologic or endoscopic residual tumor after a maximal TURBt (cT0). Survival benefits of cisplatin-based NAC were already described. The SWOG trial 3 reported a 33% reduction of estimated risk of death in the NAC plus cystectomy group compared to RC alone.

Specifically, Authors reported that survival benefit of NAC appeared to be strongly related to downstaging of the tumor to pT0: 38% and 15% in NAC plus RC and RC alone cohorts, respectively (p<0.001). At 5yr, 85% of the patients with a pT0 surgical specimen were alive. Analysis of survival according to treatment group (NAC plus cystectomy vs cystectomy alone) and pathologically free of cancer (pT0) or residual disease at the time of cystectomy evidenced comparable outcomes between groups in pT0 patients (2yr OS: 90% vs 94% in NAC plus RC and RC alone cohorts, respectively) while a slight difference occurred in patients with residual disease at the time of cystectomy (2yr OS: 66% vs 52% in NAC plus RC and RC alone cohorts, respectively). As a result, the impact of NAC seems to play a negligible role in pT0 patients, while major benefits were observed in presence of residual disease. However, all the available RCTs did not discuss the endoscopically feasibility to achieve a cT0 stage, after a maximal TURBt, prior to RC. Moreover, systematic therapies are not devoid of limitations and they need to be carefully administered, in order to reduce toxicity, to minimize the risk of cystectomy delay in patients not sensitive to chemotherapy and to reduce the impact of NAC on surgical and health related quality of life (HRQoL) outcomes. Therefore, it is necessary to improve the selection criteria of patients' candidates for NAC plus cystectomy.

The hypothesis of investigators is that performing NAC in the absence of residual disease, after a maximal TURBt, has no survival benefit over performing an early cystectomy. Whenever endoscopically feasible, the complete resection of MIBC during TURB, particularly for T2 bladder cancer, will define a condition of cT0 stage, where probably no benefits would be observed in terms of downstaging for patients receiving NAC plus RC than those undergoing an early RC alone.

ELIGIBILITY:
Inclusion Criteria:

* diagnostic TURBt with cT2-4, cN0, cM0;
* non-radiologic or endoscopic residual tumor after a maximal TURBt (cT0);
* patients eligible to curative intent, candidate to surgical treatment and/or NAC (all patients must meet all the criteria required to be able to undergo RC and/or NAC);
* ≥ 18 yrs old;
* compliants patients able to follow the study protocol and fill in EORTC quality of life questionnaires;
* patients able to provide a written informed consent for the trial

Exclusion criteria:

* anaesthesiologic contraindications to surgery;
* palliative intent;
* patients ineligible for cisplatin-combination chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the non-inferiority of radical cystectomy (RC) alone versus neoadjuvant chemotherapy plus RC on 2 years Overall Survival (OS) rates, defined as the length of time from surgery until death from any cause. | 2 years
  Overall Survival rates

SECONDARY OUTCOMES:
To compare disease free survival (DFS) rates, defined as the length of time from surgery to local disease recurrence | 6 months, 1 year, 2 years
  To evaluate early (6 months), mid-term (1 year) and long-term (2 years) DFS rates
To evaluate metastasis free survival (MFS) rates, defined as the length of time from surgery to metastasis recurrence. | 6 months, 1 year, 2 years
  To evaluate early (6 months), mid-term (1 year) and long-term (2 years) MFS rates
To evaluate recurrence free survival (RFS), rates defined as the length of time from surgery to disease recurrence. | 6 months, 1 year, 2 years
  To evaluate early (6 months), mid-term (1 year) and long-term (2 years) RFS rates
To evaluate impact of NAC on perioperative complications rate (described accordingly to Clavien Dindo classification into minor o major complications) | Within hospital stay
  To evaluate impact of NAC on perioperative complications rate within hospital stay
To evaluate impact of NAC on postoperative complications rate described accordingly to Clavien Dindo classification into minor o major complications) | 30 days, 90 days and 180 days
  To evaluate impact of NAC on postoperative complications rate at 30 days, 90 days and 180 days
To evaluate impact of NAC on readmission rates (defined as postoperative rehospitalization) | 30 days, 90 days and 180 days
  To evaluate impact of NAC on readmission rates at 30 days, 90 days and 180 days
To compare health-related quality of life (HRQoL) outcomes, using EORTC self-assessed questionnaires | 3 months, 6 months, 1 year and 2 years
  To compare health-related quality of life (HRQoL) outcomes at 3 months, 6 months, 1 year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Simone, MD, Principal Investigator — IRCCS "Regina Elena" National Cancer Institute
Locations (1):
- Riccardo Mastroianni, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stein JP, Lieskovsky G, Cote R, Groshen S, Feng AC, Boyd S, Skinner E, Bochner B, Thangathurai D, Mikhail M, Raghavan D, Skinner DG. Radical cystectomy in the treatment of invasive bladder cancer: long-term results in 1,054 patients. J Clin Oncol. 2001 Feb 1;19(3):666-75. doi: 10.1200/JCO.2001.19.3.666. PMID 11157016
- [Result] Stein JP, Skinner DG. Radical cystectomy for invasive bladder cancer: long-term results of a standard procedure. World J Urol. 2006 Aug;24(3):296-304. doi: 10.1007/s00345-006-0061-7. Epub 2006 Mar 4. PMID 16518661
- [Result] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Result] Neoadjuvant cisplatin, methotrexate, and vinblastine chemotherapy for muscle-invasive bladder cancer: a randomised controlled trial. International collaboration of trialists. Lancet. 1999 Aug 14;354(9178):533-40. PMID 10470696
- [Result] International Collaboration of Trialists; Medical Research Council Advanced Bladder Cancer Working Party (now the National Cancer Research Institute Bladder Cancer Clinical Studies Group); European Organisation for Research and Treatment of Cancer Genito-Urinary Tract Cancer Group; Australian Bladder Cancer Study Group; National Cancer Institute of Canada Clinical Trials Group; Finnbladder; Norwegian Bladder Cancer Study Group; Club Urologico Espanol de Tratamiento Oncologico Group; Griffiths G, Hall R, Sylvester R, Raghavan D, Parmar MK. International phase III trial assessing neoadjuvant cisplatin, methotrexate, and vinblastine chemotherapy for muscle-invasive bladder cancer: long-term results of the BA06 30894 trial. J Clin Oncol. 2011 Jun 1;29(16):2171-7. doi: 10.1200/JCO.2010.32.3139. Epub 2011 Apr 18. PMID 21502557
- [Result] Takata R, Katagiri T, Kanehira M, Tsunoda T, Shuin T, Miki T, Namiki M, Kohri K, Matsushita Y, Fujioka T, Nakamura Y. Predicting response to methotrexate, vinblastine, doxorubicin, and cisplatin neoadjuvant chemotherapy for bladder cancers through genome-wide gene expression profiling. Clin Cancer Res. 2005 Apr 1;11(7):2625-36. doi: 10.1158/1078-0432.CCR-04-1988. PMID 15814643
- [Result] Takata R, Katagiri T, Kanehira M, Shuin T, Miki T, Namiki M, Kohri K, Tsunoda T, Fujioka T, Nakamura Y. Validation study of the prediction system for clinical response of M-VAC neoadjuvant chemotherapy. Cancer Sci. 2007 Jan;98(1):113-7. doi: 10.1111/j.1349-7006.2006.00366.x. PMID 17116130
- [Result] Driscoll JJ, Rixe O. Overall survival: still the gold standard: why overall survival remains the definitive end point in cancer clinical trials. Cancer J. 2009 Sep-Oct;15(5):401-5. doi: 10.1097/PPO.0b013e3181bdc2e0. PMID 19826360
- [Result] Kim HS, Jeong CW, Kwak C, Kim HH, Ku JH. Disease-Free Survival at 2 and 3 Years is a Significant Early Surrogate Marker Predicting the 5-Year Overall Survival in Patients Treated with Radical Cystectomy for Urothelial Carcinoma of the Bladder: External Evaluation and Validation in a Cohort of Korean Patients. Front Oncol. 2015 Oct 29;5:246. doi: 10.3389/fonc.2015.00246. eCollection 2015. PMID 26579498
- [Result] Witjes JA, Bruins HM, Cathomas R, Comperat EM, Cowan NC, Gakis G, Hernandez V, Linares Espinos E, Lorch A, Neuzillet Y, Rouanne M, Thalmann GN, Veskimae E, Ribal MJ, van der Heijden AG. European Association of Urology Guidelines on Muscle-invasive and Metastatic Bladder Cancer: Summary of the 2020 Guidelines. Eur Urol. 2021 Jan;79(1):82-104. doi: 10.1016/j.eururo.2020.03.055. Epub 2020 Apr 29. PMID 32360052
- [Result] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542